CLINICAL TRIAL: NCT01177865
Title: Evaluating Patient Preferences for the Treatment of Localized Prostate Cancer - A Discrete Choice Experiment
Brief Title: Study of Treatment Choice in Patients With Localized Prostate Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College London Hospitals (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Health Services Research
Other Study IDs: CDR0000682206; UCL-COMPARE; EU-21055
Record Dates: First submitted 2010-08-06; First posted 2010-08-09 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2010-11

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

INTERVENTIONS:
Other: informational intervention
Other: questionnaire administration

SUMMARY:
RATIONALE: Gathering information about patients with prostate cancer may help doctors learn more about how patients choose treatment options.

PURPOSE: This study is looking at treatment choice in patients with localized prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the importance of prostate cancer treatment characteristics to men with localized prostate cancer.
* To determine to what extent men will choose the strengths and weaknesses of one treatment over a different set of strengths and weaknesses of another treatment when making a choice between them.

Secondary

* To determine the correlation between attributes that are important to men and baseline demographics, functional status, and disease risk characteristics.

OUTLINE: This is a multicenter study.

Patients complete a 'discrete choice experiment' questionnaire presenting three treatment options based on 8 aspects of treatment. Attributes relevant to men with prostate cancer (e.g., sexual health, urinary function, return to normal activities [work, gardening, sports, shopping]) that apply to surveillance, radical therapies and new minimally-invasive therapies have been selected for consideration. Baseline demographics such as age, working/retired/unemployed/household income, prostate cancer characteristics (PSA level, Gleason grade, stage), baseline functional status (genitourinary function), and final treatment choice will also be collected in order to ascertain whether there is any relationship and association between patient preferences for treatment and these baseline demographics. Individuals will be asked to choose between the three treatment profiles.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histological diagnosis of adenocarcinoma of the prostate on transrectal or transperineal template prostate biopsies

  * Clinical stage ≤ T2c N0 M0 (radiological T3a allowed)

    * Local staging imaging as per guidelines to demonstrate localized disease (e.g., MRI, CT, and/or bone scan)
  * No metastatic disease or nodal disease outside the prostate on bone scan or cross-sectional imaging
* No prior prostate surgery for cancer control (e.g., radical prostatectomy, high-intensity focused ultrasound ablation, cryosurgery, or photodynamic therapy) or other treatment for prostate cancer
* Gleason grade ≤ 7
* Serum PSA ≤ 15 ng/mL

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior radiotherapy
* No androgen suppression/hormone treatment within the previous 12 months for prostate cancer

Ages: 45 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 432 (Estimated)
Dates: Start 2010-09; Primary Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Preferences for, and trade-offs between, the attributes of pre-treatment evaluation with general anaesthetic biopsies and post-treatment frequency of biopsies
Treatment choice in respect to risks to sexual function and urinary function, return to normal activities, aim to treat the whole gland or only cancer areas or important cancer areas, retreatment rate, and mortality rate

SECONDARY OUTCOMES:
Correlation between attributes important to men and baseline demographics, functional status, and disease risk characteristics

CONTACTS AND LOCATIONS:
Overall Officials: Mark Emberton, MD, FRCS, MBBS, Principal Investigator — University College London Hospitals
Locations (1):
- University College of London Hospitals, London, England, United Kingdom